CLINICAL TRIAL: NCT02374892
Title: The CHAPTER III Study of Young Adolescents: Congenital Heart Adolescents Participating in Transition Evaluation Research
Brief Title: The CHAPTER III Study of Young Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Women and Children's Health Research Institute (WCHRI) (Unknown); Stollery Children's Hospital Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: The CHAPTER III Study
Record Dates: First submitted 2015-02-23; First posted 2015-03-02 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Heart Defects, Congenital
Keywords: Intervention; Congenital Heart Disease; Adolescent; Education; Self-management
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Adolescents will attend a single one-on-one session with a nurse. Sessions will be youth-oriented, interactive, and engaging. They will make a health passport, go over their cardiac anatomy, watch videos among other things.
  The adolescent will be given a study email address and encouraged to contact the nurse by email or text messaging with follow-up.
  Interventions: Behavioral: CHAPTER III Study Intervention
- Usual Care (No Intervention): Youth seen in the Cardiology clinic see a nurse only to measure weight, height, and blood pressure. They rely on their cardiologist for information about their heart condition. The approach and amount of time taken by each cardiologist with a youth varies.

INTERVENTIONS:
Behavioral: CHAPTER III Study Intervention — This will involve a 60 minute interaction between the adolescent and a cardiology nurse. A MyHealth passport will be created covering the name of the adolescents' cardiac condition, previous cardiac interventions, and name and purpose of the teen's medications. Potential late cardiac complications will be discussed. The adolescent and nurse will watch videos on talking to various health professionals. The adolescent will be given a study email address and encouraged to contact the nurse by email or text messaging with follow-up
  Arms: Intervention

SUMMARY:
The CHAPTER III Study (Congenital Heart Adolescents Participating in Transition Evaluation Research) is a cluster randomized controlled trial evaluating the impact of a nurse-led transition intervention in combination with usual care, versus usual care alone, on preparing adolescents with congenital heart disease (CHD) to successfully transition from pediatric to adult cardiology care. The Canadian Pediatric Society and American Academy of Pediatrics have recommended that transition interventions begin in early adolescence. Therefore, the investigators propose to conduct a nurse-led intervention that addresses the educational needs of 13-14 year olds.

DETAILED DESCRIPTION:
BACKGROUND:

The numbers of youth and young adults with congenital heart disease (CHD) is rapidly increasing, yet youth, parents, and health care providers (HCPs) are unprepared to manage the health care transition from pediatric to adult cardiology care. Both youth and parents report significant anxiety regarding the transition process. When transition is not managed well, youth may not engage with adult HCPs,which may lead to late detection of new problems,excess morbidity, and diminished quality of life.This speaks to the urgency of addressing clinical and health services research gaps, which leave affected youth, families, HCPs, and policy makers with insufficient evidence for transition program delivery.

OBJECTIVE:

The primary aim is to determine the impact of a nurse-led transition intervention in combination with usual care, compared to usual care alone, on self-management and self-advocacy skills among 13-14 year olds with moderate or complex CHD using a validated instrument. [Hypothesis: the transition intervention will result in superior self-management and self-advocacy skills compared to usual care alone]. The secondary aim is to determine knowledge of their CHD lesion [Hypothesis: the transition intervention will result in superior knowledge of the CHD lesion compared to usual care alone].

METHODS:

Study Participants

Inclusion criteria: 13-14 year olds with moderate or complex CHD (as previously defined)who are followed at the Stollery Children's Hospital (Edmonton).

Exclusion criteria: (i) less than a Grade 6 level of reading and comprehension, based on parent report; (ii) heart transplantation, as this results in distinct health challenges.

STUDY DESIGN:

Subjects will be randomized by clusters defined by week of attendance in the pediatric cardiology clinic. Because week is the unit of randomization and not the study subject, this is a cluster randomization design. We anticipate 1-2 subjects per week will be enrolled per site, i.e. the cluster size will be ≤ 2.

INTERVENTIONS:

This intervention will be conducted by a cardiology nurse who is experienced working with teens and will a one-on-one sessions approximately 60 minutes in length. Sessions will be youth-oriented, interactive, and engaging. This session will be held in conjunction with a scheduled pediatric cardiology clinic visit. This timing minimizes the study burden and is consistent with Canadian Pediatric Society recommendations that transition interventions be delivered in clinical settings. Individual sessions, in contrast to group sessions, allow the intervention content to be patient-specific. Immediately prior to the session, the RN will review the cardiology chart to familiarize them self with the cardiac history including cardiac diagnoses, names and dates of cardiac surgical procedures and cardiac catheterizations, and current cardiac medications and doses.

The one-on-one session will combine Education and an introduction of Self-Management. It will involve an introduction to transition and its importance, a discussion of confidentiality to promote trust with the RN, the creation of a MyHealth passport, review of diagram illustrating the teen's cardiac anatomy, the introduction to websites of the Sick Kids Good2Go program, and the youth-oriented YoungAndHealthy, the introduce youth-friendly written materials about risk-taking behaviours, a review of videos of good and bad interactions with a health care provider and encouragement to contact the RN at a study email address or by text messaging with follow-up questions..

STUDY PROCEDURE:

Potential study participants will be approached in the Stollery Children's Hospital Cardiology clinic. A trained project coordinator will approach subjects on both "intervention" days and "usual care" days. The nature and purpose of the study will be explained and informed consent sought from the teen's parent(s)/guardian(s).

MEASURES:

1. The TRANSITION-Q score is a Canadian created, generic self-management skills scale for use with adolescents diagnosed with a chronic health condition who are aged 12 to 18 years. The content of the scale was designed to include a range of skills that vary from those that even young adolescents should be able to do (e.g. answer a doctor's or nurse's questions) to skills that may require instruction or training (e.g. book an appointment).consists of a knowledge scale and behavior index that reports on the youths health and self-care related knowledge and behavior.
2. Knowledge of the cardiac condition will be measured with the MyHeart Scale.
3. Chart review: Descriptive data collected from the cardiology chart will be: date of birth, CHD diagnosis, names and dates of cardiac surgical procedures and cardiac catheterizations, current use of cardiac medications (Y/N), history of missed appointments (Y/N), and cardiologist's name.

Youth will complete the MyHeart Scale and the TRANSITION-Q Questionnaire in the clinic area at enrollment for the "usual care" group, and prior to intervention for the "intervention" group. Both groups will repeat the questionnaires 1 month and 6 months post enrollment.

ELIGIBILITY:
Inclusion Criteria:

(i) moderate or complex CHD (as defined by the 2001 Bethesda Guidelines) (ii) followed at the Stollery Children's Hospital

Exclusion Criteria:

(i) less than a Grade 6 level of reading and comprehension, based on parent report (ii) heart transplantation, as this results in distinct health challenges

Ages: 13 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
TRANSITION-Q Questionnaires | 6 Months
  Change in TRANSITION-Q Questionnaire score between baseline, 1 month, and 6-months post enrollment.

SECONDARY OUTCOMES:
MyHeart Scale | 6 Months
  Change in knowledge of their heart (MyHeart score) between baseline, 1 month and 6-months post enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Mackie, MD, SM, Principal Investigator — University of Alberta
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Mackie AS, Islam S, Magill-Evans J, Rankin KN, Robert C, Schuh M, Nicholas D, Vonder Muhll I, McCrindle BW, Yasui Y, Rempel GR. Healthcare transition for youth with heart disease: a clinical trial. Heart. 2014 Jul;100(14):1113-8. doi: 10.1136/heartjnl-2014-305748. Epub 2014 May 19. PMID 24842870
- [Background] Klassen AF, Grant C, Barr R, Brill H, Kraus de Camargo O, Ronen GM, Samaan MC, Mondal T, Cano SJ, Schlatman A, Tsangaris E, Athale U, Wickert N, Gorter JW. Development and validation of a generic scale for use in transition programmes to measure self-management skills in adolescents with chronic health conditions: the TRANSITION-Q. Child Care Health Dev. 2015 Jul;41(4):547-58. doi: 10.1111/cch.12207. Epub 2014 Oct 28. PMID 25351414
- [Derived] Mackie AS, Rankin KN, Yaskina M, Gingrich J, Williams E, Schuh M, Kovacs AH, McCrindle BW, Nicholas D, Rempel GR. Transition Preparation for Young Adolescents with Congenital Heart Disease: A Clinical Trial. J Pediatr. 2022 Feb;241:36-41.e2. doi: 10.1016/j.jpeds.2021.09.053. Epub 2021 Oct 4. PMID 34619115